CLINICAL TRIAL: NCT06525870
Title: Efficacy of Topical 85%Trichloroacetic Acid in the Treatment of Low-grade Squamous Intraepithelial Lesion (LSIL) After Low-grade Abnormality of Screening Test: a Randomized Controlled Trial
Brief Title: Efficacy of Topical 85% TCA in the Treatment of LSIL After Low-grade Abnormality of Screening Test: a Randomized Controlled Trial
Acronym: Trichlosil
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 136/2567
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-07

CONDITIONS: Cervical Intraepithelial Neoplasia; Trichloroacetic Acid
Keywords: CIN1; HPV; Trichloroacetic Acid; Low-grade squamous intraepithelial lesion; LSIL; Low-grade lesion
MeSH Terms: conditions — Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions | interventions — Acetic Acid

STUDY DESIGN:
Intervention Model Description: Patients then will be randomized between the two groups. Group 1 will be intervention arm and receive 85%TCA topical application at cervical lesion and transformation zone. Group 2 will be control arm and receive topical application of 3% acetic acid at cervical lesion and transformation zone in the same manner.
Who Masked: Participant
Masking Description: The treatment is unknown to the patient but the physicians will know because the different degree of cervical tissue whitening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Participants will receive 85%TCA topical application at cervical lesion and transformation zone. Application of TCA will be guided by colposcopy using a small cotton-tipped applicators and wooden end of the applicators.
  Interventions: Drug: 85%TCA topical application
- Group 2 (Placebo Comparator): Participants will receive 3% acetic acid topical application at cervical lesion and transformation zone. Application of 3% acetic acid will be guided by colposcopy using a small cotton-tipped applicators and wooden end of the applicators.
  Interventions: Drug: 3% acetic acid

INTERVENTIONS:
Drug: 85%TCA topical application — 85%TCA topical application is done at cervical lesion and transformation zone. Application of TCA will be guided by colposcopy using a small cotton-tipped applicators and wooden end of the applicators. A thin film of TCA will be applied to cover the lesion and transformation zone.
  Other Names: Group 1
  Arms: Group 1
Drug: 3% acetic acid — 3% acetic acid topical application is done at cervical lesion and transformation zone. Application will be guided by colposcopy using a small cotton-tipped applicators and wooden end of the applicators. A thin film of acetic acid will be applied to cover the lesion and transformation zone.
  Other Names: Group 2
  Arms: Group 2

SUMMARY:
To determine the efficacy and HPV clearance of an application of 85% TCA compared to placebo in the treatment of LSIL. This is a randomized, single-blind, placebo-controlled study in 44 women aged 18-65 years with histologic-proved HPV/CIN1. The study will test whether 85% TCA application will be effective treatment in LSIL. The clinical study hypothesis is that TCA application at cervical lesion and transformation zone will achieve histologic complete remission of LSIL in significantly more patients than placebo therapy. Patients will be randomized to placebo (3% acetic acid) or 85%TCA topical application at cervical lesion and transformation zone. After 3 months, cytology, colposcopy, histology, and HPV testing will be performed. The primary endpoint is treatment efficacy defined as complete histologic remission at 3 months after treatment. The secondary endpoint is HPV clearance 3 months after treatment. The protocol for the project is approved by an Institutional Review Board (IRB). Project is totally supported by a grant from Rajavithi Hospital. There is no external funding.

DETAILED DESCRIPTION:
The study aims to determine the efficacy and HPV clearance of an application of 85% TCA compared to placebo in the treatment of LSIL. This study will be conducted in women aged 18-65 years with colposcopic-biopsy proved HPV or CIN1, have low grade abnormalities of precolposcopy cervical screening. Low grade abnormalities include ASC-US+HPV positive, LSIL, HPV 16/18, persistent high-risk HPV infection. In patients referred to the colposcopy clinic with ASC-US without HPV testing, they will be eligible if the HPV testing later performed is positive for high risk type. The study will test whether 85% TCA application will be effective treatment in LSIL. The clinical study hypothesis is that TCA application at cervical lesion and transformation zone will achieve histologic complete remission of LSIL in significantly more patients than placebo therapy. A study population is a group of patients who come to gynecology clinic after the histological diagnosis of HPV/CIN I is established. After eligibility is confirmed and demographic data is collected, patients will sign informed consent, a questionnaire will be answered by them and then all patients will have evaluation at pre-intervention check which comprised cytologic test, a type-specific HPV test (if not done previously), a colposcopy colposcopic examination with 3% acetic acid. Detail of colposcopic findings will be recorded. Patients then will be randomized between the two study groups. Group 1 will be intervention arm and receive 85%TCA topical application at cervical lesion and transformation zone. Application of TCA will be guided by colposcopy using a small cotton-tipped applicators and wooden end of the applicators. A thin film of TCA will be applied to cover the lesion and transformation zone. Applying the adjacent endocervial canal and lower part of transformation zone will be cautiously managed by using the wooden stick end of the cotton-tipped applicators soaked with TCA. Protein denaturation and precipitation were confirmed by colposcopic observation of the color change to white. Group 2 will be control arm and receive topical application of 3% acetic acid at cervical lesion and transformation zone in the same manner. At the completion of the treatment, there will be 22 patients in each group. Treatment solutions will be prepared by pharmacy. The treatment is unknown to the patient but the physicians will know because the different degree of cervical tissue whitening. After interventions, the patients will be observed for 5 minutes and will be questioned regarding uncomfortable sensations using a visual analog scale from 0 to 10 (the value 0 is defined as no symptom and 10 worst symptom). Uncomfortable sensations i.e. burning or soreness will be recorded. Patients will be advised to refrain from sexual intercourse, to use sanitary pads rather than tampons, and to shower rather than to take baths for 2 weeks. The patients will be reexamined after 2 weeks following the initial visit. They will be queried about adverse events, since the last visit. Then the patients will be examined by a bivalve vaginal speculum for any evidence of incomplete healing, ulcer and infection. They will be scheduled for second follow-up visit at 3 months after the intervention. A cytologic test, a type-specific HPV test, a colposcopy including multiple guided biopsies will be performed. For the cases with no lesion upon colposcopy, four-quadrant biopsies will be performed from each quadrant of the transformation zone. Assessment of the pathological diagnosis will be done as blindness by pathologists at 3 months after the intervention. The primary endpoint is treatment efficacy defined as complete histologic remission at 3 months after treatment. The secondary endpoint is type-specific HPV clearance at 3 months after treatment. A histologic complete remission (histologic cure) is defined as biopsy-proved normal histology at the time of final colposcopy examination at 3-month follow-up. Because all of patients in this study have low-grade histology, a histologic regression will be defined as biopsy-proved normal histology at the time of final colposcopy examination as well. A histologic progression is defined as CIN2 or worse lesions that are demonstrated on biopsy and histologic persistence is defined as HPV/CIN 1 lesions that are again demonstrated on biopsy at the final colposcopy examination. To determine the sample size, a randomized clinical trial sample size formula where type one (α) error was considered as 5% and the study power as 80% is used. Based on previous studies and considering 46.6% as the difference in complete remission between the two groups. A sample size of 17 patients in each group is needed (α=0.05, power=0.8). Allowing for a dropout rate of 20%, the final sample size is determined to be 22 subjects per group. The total sample size is 44. The analyses will be conducted in all randomized subjects according to the intention-to-treat (ITT) principle. Patients with missing data on remission or regression of LSIL and HPV clearance resulting from refusal to continue participation, and those who failed to appear at scheduled follow-up visits, is regarded as nonresponders. Continuous variables will be summarized by descriptive statistics, including number, mean, median, standard deviation, minimum, and maximum. Categorical variables will be summarized by number and percentage. Independent samples Student's t test to detect mean differences in baseline measures as well as interventions between the two groups. In addition, paired samples t-test is used to detect within-group differences. Pearson Chi-square test is used for comparison of categorical variables. The protocol for the project receives ethics approval from the Institutional Review Board and it is supported by a grant from Rajavithi Hospital. There is no external funding.

ELIGIBILITY:
Inclusion criteria

* Women, 18-65 years of age, colposcopic biopsy confirmed CIN1 or HPV (LSIL) preceded by low-grade cervical screening test, i.e. ASCUS HPV positive, LSIL, HPV 16/18 positive, persistent high-risk HPV infection.
* Willing to participate in this trial

Exclusion criteria

* Women diagnosed with previous or concurrent invasive carcinoma of the cervix
* Women with history of pelvic radiotherapy
* Pregnant women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete histologic remission at 3 months | 3 months
  Complete remission (histologic cure) is defined as biopsy-proved normal histology at the time of final colposcopy/biopsy examination at 3-month follow-up.

SECONDARY OUTCOMES:
Type-specific HPV clearance at 3 months after treatment | 3 months
  Defined as previous type-specific HPV positivity at the initilal assesement become negative at follow-up reassessment visit

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Thailand, Bangkok, Thailand